CLINICAL TRIAL: NCT00315393
Title: Determining Disease Activity Biomarkers in Individuals With Granulomatosis With Polyangiitis (Wegener's) and Microscopic Polyangiitis
Brief Title: Longitudinal Protocol for Granulomatosis With Polyangiitis (Wegener's) and Microscopic Polyangiitis
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Other Study IDs: VCRC5505; U54AR057319 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis; Wegener's
Keywords: GPA; MPA; WG
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum and plasma), urine, and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Granulomatosis with polyangiitis (Wegener's) (GPA) and microscopic polyangiitis (MPA) are two rare immune system disorders that cause the inflammation of blood vessels, or vasculitis. In order to properly treat these diseases, it is critical that the level of disease activity can be determined over the course of the disease. The purpose of this study is to determine new biological markers, or biomarkers, that may be used to assess the severity of disease in people with GPA or MPA.

DETAILED DESCRIPTION:
GPA and MPA are two autoimmune disorders that cause systemic vasculitis. GPA commonly affects the upper respiratory tract, the lungs, and the kidneys. MPA is marked by kidney inflammation, weight loss, skin lesions, nerve damage, and fever. Many patients with WG or MPA show no visible symptoms of active disease; it is known that underlying subclinical disease activity leads to long-term damage in these patients. Also, because it is difficult to monitor WG and MPA disease activity, it is difficult for clinicians to know when and how to treat these patients. This study will use new scientific methods to identify new biomarkers that can be used to monitor disease activity in GPA and MPA patients. These biomarkers may be used to help direct clinical care for GPA and MPA patients and assist in future drug development.

Study visits will occur monthly for the first year, then every 3 months thereafter for the remainder of the study. Blood and urine collection will occur at every visit. A physical exam and medical and medication history will occur every 3 months; also, participants will be asked to complete several questionnaires to assess disease activity, health status, and tobacco, alcohol, and drug use. Participants may have additional study visits if a disease flare or disease-related complications occur during the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GPA or MPA. Widely accepted diagnostic criteria, as opposed to classification criteria or definitions, have not been developed for GPA and MPA.
* For diagnosis of GPA, meets at least 2 of the following 5 modified American College of Rheumatology (ACR) criteria:

  1. Nasal or oral inflammation with oral ulcers or nasal discharge with pus or blood
  2. Abnormal chest radiograph with nodules, fixed infiltrates, or cavities
  3. Urinary sediment with microhematuria or red cell casts
  4. Granulomatous inflammation within the wall of an artery or in the perivascular area on biopsy
  5. Antineutrophil cytoplasmic antibody (ANCA) positive by enzyme immunoassay for either PR3- or MPO-ANCA
* For diagnosis of MPA, meets the Chapel Hill Consensus Conference Definition for MPA:

  1. Necrotizing vasculitis, with few or no immune deposits, that affects small vessels (i.e., capillaries, venules, arterioles)
  2. Necrotizing arteritis involving small- and medium-sized arteries may be present
  3. Necrotizing glomerulonephritis is very common
  4. Pulmonary capillaritis often occurs
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Simultaneous diagnoses of both GPA and MPA
* Granulomatosis with polyangiitis (Churg-Strauss)
* Takayasu's arteritis
* Giant cell arteritis
* Polyarteritis nodosa
* Cogan's syndrome
* Behcet's disease
* Sarcoidosis
* Kawasaki disease
* Tuberculosis or any atypical mycobacterial infections
* Deep fungal infections
* Lymphoma, lymphomatoid granulomatosis, or any other type of cancer that mimics anti-neutrophil cytoplasmic antibody-associated vasculitis (AAVs)
* Cryoglobulinemic vasculitis
* Systemic lupus erythematosus
* Rheumatoid arthritis
* Mixed connective tissue disease or any overlapping autoimmune syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with granulomatosis with polyangiitis (Wegener's)and microscopic polyangiitis. Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 1046 (Actual)
Dates: Start 2006-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Discover biomarkers in GPA/MPA capable of measuring disease activity and response to treatment. | Study completion

SECONDARY OUTCOMES:
Measure the predictive value of biomarkers for clinical outcome in GPA/MPA | Study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (8):
- United States (6):
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Background] Borgmann S, Haubitz M. Genetic impact of pathogenesis and prognosis of ANCA-associated vasculitides. Clin Exp Rheumatol. 2004;22(6 Suppl 36):S79-86. PMID 15675141
- [Background] Cooley P, Taylor KH, Czika W, Seifer C, Taylor JF. Analysis of a biomarker for Wegener's granulomatosis. Int J Immunogenet. 2005 Aug;32(4):237-43. doi: 10.1111/j.1744-313X.2005.00519.x. PMID 16026591
- [Background] Jagiello P, Gross WL, Epplen JT. Complex genetics of Wegener granulomatosis. Autoimmun Rev. 2005 Jan;4(1):42-7. doi: 10.1016/j.autrev.2004.06.003. PMID 15652778
- [Background] Radice A, Sinico RA. Antineutrophil cytoplasmic antibodies (ANCA). Autoimmunity. 2005 Feb;38(1):93-103. doi: 10.1080/08916930400022673. PMID 15804710
- [Background] Stone JH, Rajapakse VN, Hoffman GS, Specks U, Merkel PA, Spiera RF, Davis JC, St Clair EW, McCune J, Ross S, Hitt BA, Veenstra TD, Conrads TP, Liotta LA, Petricoin EF 3rd; Wegener's Granulomatosis Etanercept Trial Research Group. A serum proteomic approach to gauging the state of remission in Wegener's granulomatosis. Arthritis Rheum. 2005 Mar;52(3):902-10. doi: 10.1002/art.20938. PMID 15751091
- [Derived] Tomasson G, Boers M, Walsh M, LaValley M, Cuthbertson D, Carette S, Davis JC, Hoffman GS, Khalidi NA, Langford CA, McAlear CA, McCune WJ, Monach PA, Seo P, Specks U, Spiera R, St Clair EW, Stone JH, Ytterberg SR, Merkel PA. Assessment of health-related quality of life as an outcome measure in granulomatosis with polyangiitis (Wegener's). Arthritis Care Res (Hoboken). 2012 Feb;64(2):273-9. doi: 10.1002/acr.20649. PMID 21954229
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/cms/vcrc/
- See also: Rare Diseases Clinical Research Consortium — http://rarediseasesnetwork.org/